CLINICAL TRIAL: NCT06304857
Title: A Multicentre, Randomised, Double-blind, Placebo-controlled Phase III Study, Evaluating the Effect of Dapagliflozin on Prevention of Cardiotoxicity in Breast Cancer Patients Undergoing Anthracycline-based Chemotherapy
Brief Title: CardioPROTECTion with Dapagliflozin in Breast Cancer Patients Treated with AnthrAcycline - PROTECTAA TRIAL
Acronym: PROTECTAA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: 4th Military Clinical Hospital with Polyclinic, Poland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2022/ABM/01/00039; 2023-506631-15-00 (Other: EUCT)
Record Dates: First submitted 2023-10-09; First posted 2024-03-12 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer; Heart Failure
Keywords: breast cancer; heart failure; ejection fraction; anthracyclines
MeSH Terms: conditions — Breast Neoplasms; Heart Failure | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dapagliflozin (Experimental): Dapagliflozin 10 mg tablet orally once daily for 12 months
  Interventions: Drug: Dapagliflozin
- Placebo (Placebo Comparator): Placebo tablet matching dapagliflozin orally once daily for 12 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin — 10 mg tablet q.d
  Other Names: Farxiga; Forxiga
  Arms: Dapagliflozin
Drug: Placebo — tablet matching dapagliflozin 10 mg q.d
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of dapagliflozin on the incidence of cancer therapeutics-related cardiac dysfunction in patients with breast cancer receiving anthracycline treatment.

DETAILED DESCRIPTION:
This is a multicentre, randomised, double-blind, placebo-controlled phase III study, evaluating the effect of dapagliflozin versus placebo on prevention of cardiotoxicity in breast cancer patients undergoing anthracycline-based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years and < 80 years.
* Diagnosis of invasive breast cancer [stage I-III] and planned anthracycline treatment within 60 days.
* Signed Informed Consent to participate in the study.

Exclusion Criteria:

* Urinary tract infection with the need for treatment with an antibiotic 48 hours before the scheduled start of anthracycline treatment.
* Recognised heart failure or symptoms which, in the opinion of the investigator may be a symptom of undiagnosed heart failure.
* Left ventricular ejection fraction < 50% at the time of the screening.
* Severe valvular heart disease.
* A history of clinically significant arrhythmia, including atrial fibrillation regardless of type (at discretion of the investigator).
* A history of stroke.
* Cardiomyopathy: congenital, post-inflammatory, toxic, infiltrative (e.g. amyloidosis, sarcoidosis, haemochromatosis), postnatal or hypertrophic.
* Pulmonary hypertension.
* Uncontrolled arterial pressure or systolic pressure < 80 mmHg at screening (at the discretion of the investigator).
* BMI > 40 kg/m2.
* Diagnosed type 1 or type 2 diabetes or fasting glucose ≥ 126 mg/dl or HbA1C ≥ 6,5% (48 mmol/mol).
* Pregnancy or breastfeeding.
* Lack of compliance to use highly effective method of birth control.
* Expected or possible treatment with epirubicin or liposomal doxorubicin within 12 months.
* Taking another study drug or drugs from the group of SGLT2 inhibitors up to 6 months before the screening visit.
* Taking semaglutide, liraglutide and metformin during the 30 days preceding the screening visit.
* eGFR < 25 ml/min/1.73m2 according to CKD EPI.
* Life expectancy < 12 months or cancer disease stage IV according to the TNM classification.
* Alanine transaminase or aspartate transaminase levels above 2.5 times the local norm.
* Anemia with Hemoglobin < 9 g/dl.
* Kidney failure > G2 (according to KDIGO classification).
* Liver disorders, Child-Pugh score > 4.
* Known, active infections with HIV, HBV, HCV, tuberculosis.
* Any other condition which, in the opinion of the investigator, makes it impossible to fulfill the requirements for participation in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary efficacy composite endpoint (cancer therapeutics related cardiac dysfunction) at 12 months. | 12 months
  Incidence of cancer therapeutics related cardiac dysfunction defined as:
  1. the appearance of heart failure symptoms (NYHA class I-IV) due to an impairment of heart function or structure within 12 months; or
  2. asymptomatic decrease in left ventricular ejection fraction > 10% after 12 months; or
  3. asymptomatic decrease in left ventricular ejection fraction < 10% but up to 40-49% after 12 months; or
  4. asymptomatic decrease in global left ventricular longitudinal strain >15% after 12 months; or
  5. asymptomatic increase in biomarkers (troponin I > upper reference limit (99th centile) and increase of at least 30% from pre-treatment concentration or NTproBNP > 125 pg/ml and increase of at least 30% from baseline) after 12 months.

SECONDARY OUTCOMES:
Secondary efficacy composite endpoint (cancer therapeutics related cardiac dysfunction) at 6 months. | 6 months
  Incidence of cancer therapeutics related cardiac dysfunction defined as:
  1. emergence of heart failure symptoms (NYHA class I-IV) due to impaired cardiac function or structure at 6 months; or
  2. decrease LVEF > 10% after 6 months; or
  3. decrease LVEF < 10% but to a value of 40-49% after 6 months; or
  4. a decrease in global longitudinal strain of > 15% after 6 months; or
  5. asymptomatic increase in biomarkers (troponin I > upper reference limit (99th centile) and an increase of at least 30% from pre-treatment concentration or NTproBNP >125pg/ml and an increase of at least 30% from baseline) after 6 months.
Change in left ventricular ejection fraction at 6 and 12 months. | 6 and 12 months
  Assessed by transthoracic echocardiography.
Change in left ventricular diastolic function at 6 and 12 months. | 6 and 12 months
  Assessed as the ratio of E/E', i.e. maximum mitral annular inflow velocity during the rapid ventricular filling phase, to maximum mitral annular motion velocity by tissue Doppler during the rapid ventricular filling phase.
Change in Troponin I after 6 and 12 months. | 6 and 12 months
  Secondary.
Change in NTproBNP levels at 6 and 12 months. | 6 and 12 months
  Secondary.
Quality of life at 6 and 12 months assessed using the five-dimensional EQ-5D questionnaire. | 6 and 12 months
  The EQ-5D questionnaire consists of two parts: descriptive one, which measures five dimensions of health (mobility, self care, usual activities, pain & discomfort, anxiety & depression) and EQ Visual Analogue Scale numbered from 0 to 100, where higher value indicate better self-reported health.
Occurrence of death from any cause. | 13 months (additional 1 month of safety follow-up after end of treatment).
  Secondary safety endpoint.
Composite endpoint of cardiovascular events. | 13 months (additional 1 month of safety follow-up after end of treatment).
  Secondary safety endpoint. Occurrence of death from cardiovascular causes, nonfatal myocardial infarction, non-fatal stroke.
Occurrence of death from any cardiovascular reasons. | 13 months (additional 1 month of safety follow-up after end of treatment).
  Secondary safety endpoint.
Occurrence of non-fatal myocardial infarction. | 13 months (additional 1 month of safety follow-up after end of treatment).
  Secondary safety endpoint.
Occurrence of non-fatal stroke. | 13 months (additional 1 month of safety follow-up after end of treatment).
  Secondary safety endpoint.
Occurrence of hypoglycaemia. | 13 months (additional 1 month of safety follow-up after end of treatment).
  Secondary safety endpoint. Hypoglycaemia is defined as serum glucose level 3 mmol/l (<54 mg/dl) with coexisting related clinical symptoms.
Occurrence of ionic disorders. | 13 months (additional 1 month of safety follow-up after end of treatment).
  Secondary safety endpoint, defined as occurrence of:
  * Sodium plasma level of >150 mmol/L
  * Potassium plasma level of >6.0 mmol/L
Occurrence of renal failure. | 13 months (additional 1 month of safety follow-up after end of treatment).
  Secondary safety endpoint. Defined as:
  * sustained (i.e. >28 days) decline in eGFR ≥50% AND/OR
  * reaching end stage renal disease defined as:
    * sustained (i.e. >28 days) eGFR <15 mL/min/1.73 m2
    * chronic dialysis treatment
    * receiving a renal transplant AND/OR
  * renal death
Occurrence of hypersensitivity to investigated drug. | 13 months (additional 1 month of safety follow-up after end of treatment).
  Secondary safety endpoint. Any unexpected adverse drug reaction (UADR).
Occurrence of allergic reactions. | 13 months (additional 1 month of safety follow-up after end of treatment).
  Secondary safety endpoint. Any hypersensitivity reaction with proven immunological pathomechanism (types I-IV according to Coombs and Gell).
Occurrence of infection. | 13 months (additional 1 month of safety follow-up after end of treatment).
  Secondary safety endpoint. Any symptomatic infection (viral, bacterial or fungal).

CONTACTS AND LOCATIONS:
Overall Officials: Waldemar Banasiak, PhD, MD, Principal Investigator — 4th Military Clinical Hospital with Polyclinic
Locations (3):
- Poland (3):
  - 4th Military Clinical Hospital with Polyclinic, Wroclaw, Lower Silesian Voivodeship
  - Lower Silesian Centre for Oncology, Lung Diseases and Hematology, Wroclaw, Lower Silesian Voivodeship
  - Military Medical Institute, Warsaw, Masovian Voivodeship

IPD SHARING:
Plan to Share IPD: No